CLINICAL TRIAL: NCT06131138
Title: Effects of Aquatic Exercises and Core Strengthening on Disability, Flexibility and Postural Stability in Weightlifters With Chronic Low Back Pain.
Brief Title: Aquatic Exercises VS Core Strengthening on Disability, Flexibility and Postural Stability in Weightlifters.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0440
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Hydrotherapy; Core Stability; Resistance Training; Low Back Pain
Keywords: Aquatic exercises; Core strengthening; Weightlifters; chronic low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Randomized clinical trials
Who Masked: Outcomes Assessor
Masking Description: The assessor who will take the readings is blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquatic exercises (Experimental): Group A will perform aquatic exercises that includes abdominal hollowing, vertical downward press, lateral downard press, straight leg raising, trading water and deep water running. Three sessions per week for 6 weeks.
  Interventions: Other: Aquatic exercises
- Core strengthening (Experimental): Group B will perform core strengthening exercises that includes abdominal hollowing, side bridge, spine extension bridge, straight leg raise from prone, alternate arm and leg raise from quadruped and prone bridge. Three sessions per week for 6 weeks
  Interventions: Other: Core strengthening

INTERVENTIONS:
Other: Aquatic exercises — This include aquatic exercises thrice as week for 6 weeks.
  Arms: Aquatic exercises
Other: Core strengthening — This include core strengthening exercises thrice a week for 6 weeks
  Arms: Core strengthening

SUMMARY:
The study is randomized and single blinded.Ethical approval is taken from ethical committee of Riphah international university, Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A and group B through sealed envelope method by non probability convenient random sampling technique. Subjects in group A will receive aquatic exercises. Group B will receive core strengthening.

DETAILED DESCRIPTION:
The objective of the study is to determine the effects of aquatic exercises verses core strengthening on disability, flexibility and postural stability in weightlifters with chronic low back pain. The study is randomized and single blinded. Ethical approval is taken from ethical committee of Riphah international university Lahore. Participants who meet the inclusion criteria will be enrolled and allocated in group A and group B through sealed envelope method by non probability convenient random sampling technique. subjects in group A will receive Aquatic exercises. Group B will receive Core strengthening. The outcome measures will be assessed by modified Oswestry Low back disability index , Modified finger_tip to floor method and New York Posture Rating Chart. The data will be analyzed by SPSS, Version 25. Statistical significance is P=0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age of participants between 20-35 years
* Experienced male weightlifters from past 6 months to in practice.
* Participants must have chronic low back pain for at least three months before enrollin

Exclusion Criteria:

* Patients with significant back pain who need rapid medical or surgical treatment.
* History of respiratory or heart diseases
* Water related anxiety or inability to adapt to aquatic environment.
* Participants with prior back surgery i.e. had surgery within six months.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
Disability | Pre and 6 week post international
  Disability will be measured by modified Oswestry Low back disability index.
Flexibility | Pre and 6 weeks post interventional
  Flexibility will be measured by modified Finger_tip to floor method.
Postural stability | Pre and 6 weeks post interventional
  Postural stability will be measured by New York Posture Rating Chart

CONTACTS AND LOCATIONS:
Overall Officials: Laraib Iqbal, DPT, Principal Investigator — Study principal investigator
Locations (1):
- Firehouse fitness gym, Sargodha, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu F, Zhang M, Wang D, Hong Q, Zeng C, Chen W. Yoga compared to non-exercise or physical therapy exercise on pain, disability, and quality of life for patients with chronic low back pain: A systematic review and meta-analysis of randomized controlled trials. PLoS One. 2020 Sep 1;15(9):e0238544. doi: 10.1371/journal.pone.0238544. eCollection 2020. PMID 32870936
- [Background] Tagliaferri SD, Miller CT, Owen PJ, Mitchell UH, Brisby H, Fitzgibbon B, Masse-Alarie H, Van Oosterwijck J, Belavy DL. Domains of Chronic Low Back Pain and Assessing Treatment Effectiveness: A Clinical Perspective. Pain Pract. 2020 Feb;20(2):211-225. doi: 10.1111/papr.12846. Epub 2019 Nov 11. PMID 31610090
- [Background] Grabovac I, Dorner TE. Association between low back pain and various everyday performances : Activities of daily living, ability to work and sexual function. Wien Klin Wochenschr. 2019 Nov;131(21-22):541-549. doi: 10.1007/s00508-019-01542-7. Epub 2019 Sep 6. PMID 31493101
- [Background] Abadi FH, Sankaravel M, Zainuddin FF, Elumalai G, Razli AI. The effect of aquatic exercise program on low-back pain disability in obese women. J Exerc Rehabil. 2019 Dec 31;15(6):855-860. doi: 10.12965/jer.1938688.344. eCollection 2019 Dec. PMID 31938709
- [Background] Hlaing SS, Puntumetakul R, Khine EE, Boucaut R. Effects of core stabilization exercise and strengthening exercise on proprioception, balance, muscle thickness and pain related outcomes in patients with subacute nonspecific low back pain: a randomized controlled trial. BMC Musculoskelet Disord. 2021 Nov 30;22(1):998. doi: 10.1186/s12891-021-04858-6. PMID 34847915